Protocol number: VAR-2021-03

# Varian ProBeam Proton Therapy System China Clinical Trial (Hefei).

(Prospective, two-centered, single- group target value method)

| Name of the medical device for investigation | Proton therapy system | |
|---|---|---|
| Model | ProBeam | |
| Management categories for investigational medical devices | Class III medical devices | |
| Class III medical devices clinical trial approval | subject to Yes□ No☑ | |
| Similar products in China | | Yes□ No☑ |
| Protocol version number and date | Version number: 1 4, Version date: 2022.06 | |
| Clinical trial institutions | Anhui Provincial Hospital | |
| researcher | Zhang Hongyan | |
| Sponsor | Varian Medical Systems Trading (Beijing)<br>Co., Ltd | |
| agent | NA | |

#### **Privacy Statement**

All information in this scheme is owned byOwned by the sponsor, only for the investigator and its authorized personnel, institutional medical device clinical trial management department, institutional ethics committee and supervision and management department and other relevant personnel for review. It is strictly forbidden to disclose any information to third parties unrelated to this study without the sponsor's written permission, except for the necessary explanation when signing the informed consent form with the subject of this study.

## **Directory**

| List of abbreviations | 3 |
|------------------------------------------------------------|---------------|
| Protocol summary | 7 |
| 1 Sponsor information | 13 |
| 1.1 Name of the sponsor | 13 |
| 1.2 Sponsor address | 13 |
| 1.3 The name, address, contact information and relevant | qualification |
| documents of the agent | 13 |
| 2 Purpose and content of clinical trial | 13 |
| 2.1 Objective | 13 |
| 2.2 content | 14 |
| 3 Overall design | 15 |
| 3.1 Trial design | 15 |
| 4 Statistical considerations | 33 |
| 4.1 Statistical design, methods, and analytical protocols | 33 |
| 4.2 Sample size calculation | 33 |
| 4.3 The level of significance and power of clinical trials | 34 |
| 4.4 Expected shedding rate | 34 |

| 4.5 Criteria for passing/failing clinical trial results |
|---|
| 4.6 Criteria and reasons for terminating trials on statistical grounds35 |
| 4.7 Statistical methods of data, together with methods of dealing with |
| missing, unused or erroneous data and irrational data35 |
| 4.8 Procedures for reporting deviations from the original statistical plan38 |
| 4.9 Selection criteria and rationale for participants included in the analysis |
| 38 |
| 4.10 Covariate and subgroup analysis |

### List of abbreviations

| Abbreviatio ns | Full spelling in English | Chinese translation |
|---|---|---|
| 3DCRT | 3-Dimensional Conformal Radiation Therapy | 3D conformal radiation therapy |
| ADL | Activities of Daily Living | Daily activities |
| AE | Adverse Events | Bad Incident |
| WHITE | Serum Albumin | Serum albumin |
| OLD | Alanine Aminotransferase | Alanine aminotransferase |
| APTT | Activated Partial Thromboplastin Time | Activation of partial thromboplastin time |
| AST | Aspartate Aminotransferase | Glutamate aminotransferase |
| GOOD | Blood Urea Nitrogen | Urea nitrogen |
| Ccr | Endogenous Creatinine Clearance Rate | Creatinine clearance |
| CFDA | China Food and Drug Administration | State Food and Drug Administration |
| СН | Chordoma | Chordoma |
| CK-MB | Creatine Kinase Isoenzymes-MB | Creatine kinase isoenzymes |
| СР | Child-Pugh | - |
| CR | Complete Response | Complete remission |
| CRA | Clinical Research Associate | Clinical monitor |
| CRF | Case Report Form | Case report form |
| CTCAE | Common Terminology Criteria for Adverse<br>Events | Common terminology criteria for adverse events |
| cTn | Cardiac Troponin | Troponin |
| CTV | Clinical Target Volume | Clinical targets |
| DART | Dynamic Adaptive Radiation Therapy | Dynamically adapted radiotherapy techniques |
| DIPS | Digital Imaging Positioning System | Digital image positioning system |
| DOR | Duration of Response | Duration of mitigation |
| DRR | Digitally Reconstruction Radiograph | Digitally reconstructed radiography |
| DVH | Dose Volume Histogram | Volume dose histogram |
| EC | Ethics Committee | Ethics Committee |
| ECOG | Eastern Cooperative Oncology Group | Eastern U.S. Oncology Collaborative<br>Group |
| eCRF | Electronic Case Report Form | Electronic case report form |

| Abbreviatio<br>ns | Full spelling in English | Chinese translation |
|---|---|---|
| EDC | Electronic Data Capture System | Electronic data collection systems |
| ERA | Erythrocyte | Urine red blood cell count |
| FAS | Full Analysis Set | Full analysis set |
| FPG | Fasting Plasma Glucose | Fasting blood sugar |
| GCP | Good Clinical Practice | Good Clinical Trial Management<br>Practice for Medical Devices |
| GLU | Glucose | Urine sugar |
| GTV | Gross Tumor Volume | Gross tumor area |
| HBV | Hepatitis Virus B | Hepatitis B virus |
| HCG | Human Chorionic Gonadotropin | Blood pregnancy test |
| HCV | Hepatitis Virus C | Hepatitis C virus |
| HGB | Hemoglobin | haemoglobin |
| HIV | Human Immunodeficiency Virus | Human immunodeficiency virus |
| ICF | Informed Consent Form | Informed consent |
| IGRT | Image-Guided Radiation Therapy | Image-guided radiation therapy |
| IMPT | Intensity Modulated Proton Therapy | Conformal intensity-modulated proton therapy |
| IMRT | Intensity Modulated Radiation Therapy | Conformal intensity-modulated radiation therapy |
| INR | International Normalized Ratio | International standardized ratio |
| LET | Linear Energy Transfer | Linear energy transfer |
| LEU | Leucocyte | Urine white blood cell count |
| LGG | Low-Grade Glioma | Low-grade glioma |
| LVEF | Left Ventricular Ejection Fractions | Left ventricular ejection fraction |
| Mb | Myoglobin | myoglobin |
| NEUT | Neutrophil | Neutrophils |
| NMPA | National Medical Products Administration | State Drug Administration |
| NPC | Nasopharyngeal Carcinoma | Nasopharyngeal carcinoma |
| NSCLC | Non-Small-Cell Lung Cancer | Non-small cell lung cancer |
| NYHA | New York Heart Association | New York Heart Society |
| OAR | Organ at Risk | Endangers organs |

| Abbreviatio ns | Full spelling in English | Chinese translation |
|---|---|---|
| WHETHER | Occult Blood Test | Occult blood test |
| OIS | Oncology Information System | Radiation therapy management software |
| OPC | Oropharyngeal Cancer | Oropharyngeal cancer |
| ORR | Objective Response Rate | Objective response rate |
| THE | Overall Survival | Overall lifetime |
| PBS | Pencil Beam Scanning | Pen beam scanning |
| PD | Progressive Disease | Disease progression |
| PFS | Progression-free Survival | Progression-free survival |
| PLT | Platelet | platelet |
| PPS | Per-Protocol Set | Conforms to the scenario set |
| PR | Partial Response | Partial remission |
| FOR | Protein | Urine protein |
| PRV | Planning Organ-at-Risk Volume | Plan to endanger organs |
| PSA | Prostate Specific Antigen | Prostate-specific antigen |
| PSI | Paul Scherrer Institute | Paul Scheller Institute, Switzerland |
| PT | Prothrombin Time | Prothrombin time |
| PTC | Proton Treatment Console | Proton therapy console |
| PTV | Planning Target Volume | Plan the target |
| QA | Quality Assurance | quality assurance |
| QOL | Quality-of-Life | Quality of life assessment |
| RBC | Red Blood Cell | erythrocyte |
| RBE | Relative Biological Effectiveness | Relative biological effects |
| RECIST 1.1 | Response Evaluation Criteria in Solid Tumors<br>RECIST Version 1.1 | Tumor efficacy evaluation criteria version 1.1 |
| RVR | Remaining Volume at Risk | Remaining danger areas |
| SAE | Serious Adverse Events | Serious adverse events |
| SBRT | Stereotactic Body Radiation Therapy | Stereotactic radiosurgery |
| SCIC | Second Channel Integrity Check | Second integrity check |
| SCLC | Small Cell Lung Cancer | Small cell lung cancer |

| Abbreviatio<br>ns | Full spelling in English | Chinese translation |
|---|---|---|
| Scr | Serum Creatinine | creatinine |
| SD | Stable Disease | The disease is stable |
| SDV | Source Data Validation | Raw data verification |
| SLD | Sum of Longest Diameter | The sum of the longest diameters of the tumor |
| SOBP | Spread-out Bragg Peak | Extend Bragg Peak |
| SOP | Standard Operating Procedure | Standard operating procedures |
| SS | Safety Set | Security datasets |
| ETC | Serum Total Bilirubin | Total serum bilirubin |
| TV | Treated Volume | Treatment area |
| ULN | Upper Limit of Normal | Upper limit of normal value |
| VMAT | Volumetric-Modulated Arc Therapy | Volumetric rotational intensity-<br>modulated radiotherapy |
| WBC | White Blood Cell | white blood cell |
| WHO | World Health Organization | World Health Organization |

## **Protocol summary**

| | · |
|---|---|
| The name of | |
| the | Varian ProBeam Proton Therapy System China Clinical Trial (Hefei). |
| experiment | varian 11020am 110ton 1110tapy System China China (110101). |
| | Investigational medical device: proton therapy system (hereinafter referred to as |
| Device name | ProBeam). |
| Manage | Class III (classification: 05 radiotherapy equipment01 radiotherapy equipment02 |
| categories | medical light ion therapy system). |
| Scope of | Proton therapy system provide precision radiation therapy protons for lesions, tumors, |
| application | and conditions in the patient's body that require radiation therapy. |
| Scope of the | Cancer patients, including tumors of the nervous system, head and neck, chest, |
| test | abdomen, spine, pelvis, limbs, etc |
| Trial design | Prospective, two-centered, single-group target value method |
| | Clinical trial (screening-short-term follow-up): The data obtained by using Proton Beam |
| Tr. dal and a | system (ProBeam) for radiation therapy in tumor patients compared with the target value |
| Trial and | to evaluate the effectiveness and safety of ProBeam for radiation therapy in tumor |
| long-term | patients to provide clinical basis for product registration application. |
| follow-up | Long-term follow-up: The long-term efficacy and safety of ProBeam for radiation |
| purposes | therapy in cancer patients were evaluated by using the long-term follow-up data of |
| | ProBeam for radiation therapy in cancer patients. |
| | 47 cases. |
| | Among them, the number of head and neck, chest, abdomen, spine and pelvic tumors |
| Sample size | is distributed as evenly as possible. |
| | Intensity modulated Proton Therapy (IMPT) technology and respiratory gating |
| | technology should be used and verified in this study. |
| clinical trial | |
| Number of | 2 |
| institutions | |
| | The screening period from signing the informed consent form to enrollment is |
| The expected | expected to be 4 weeks, the treatment period is 1~8 weeks, and the short-term |
| duration of | follow-up and long-term follow-up after the last treatment are divided into |
| the | short-term follow-up and long-term follow-up, and the maximum duration |
| participant's | of expected participation of each subject from screening to the end of short-term |
| participation | follow-up is 12 weeks +3 months. Long-term follow-up continued after the end of the |
| | short-term follow-up until the fifth year after the end of the last radiotherapy. |
| Expected | The first subject is expected to be enrolled in December 2021, and the clinical trial |
| overall | institution expects to enroll 8-18 subjects per month, for a total enrollment time of |
| duration of | about 4 months, and the last 1 subject ends the trial (short-term follow-up) is End In |
| clinical trials | September 2022, the overall duration of the clinical trial included all working |
| and long-term | hours before, during and after the start of all clinical trials, and the overall duration of |
| follow-up | the clinical trial was 16 months. |

| | The first subject is expected to start long-term follow-up in May 2022 and the last |
|---|---|
| | one subject to end long-term follow-up in June 2027, and the overall duration |
| | of long-term follow-up in clinical trials includes all clinical runs, After all working |
| | hours ended, the total long-term follow-up period for clinical studies was |
| | approximately 62 months. |
| | Disease Control Rate (DCR). |
| | Evaluation time: 3 months $\pm 7$ days after the last treatment. |
| | Definition of indicators: Complete Response (CR), Partial Response (PR), Stable |
| | Disease (SD) for disease control; No biochemical recurrence at the end of prostate |
| Primary | cancer treatment, no regional lymph nodes or distant metastases, considered disease |
| effectiveness | control. Proportion of participants who developed disease control three months after |
| <b>Evaluation</b> | the end of the last radiotherapy. Participants who discontinued the trial for any reason |
| indicators | (except loss to follow-up) before the end of radiation therapy were considered to have |
| indicators | progression (PD) or uncontrolled. |
| | Evaluation methodology: Response Evaluation Criteria in Solid Tumors RECIST |
| | Version 1.1 (RECIST 1.1) by an independent imaging review team Changes in |
| | tumour CT or MRI imaging before and after treatment were assessed. At 3 months |
| | of radiographic evaluation, if PD is found, PET-CT is required to confirm it. |
| | (1) Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 toxicity |
| | ratio |
| | Evaluation time: 3 months $\pm$ 7 days after the end of the last treatment. |
| | Indicator definition: Proportion of subjects with grade 3 toxicity during the |
| The main | trial cycle. |
| safety | Evaluation methodology: Investigators recorded AEs that occurred during the |
| evaluation | clinical trial cycle and graded them according to CTCAE V5.0. |
| index | (2) CTCAE grade 4 and 5 toxicity ratio |
| mucx | Evaluation time: the entire clinical trial cycle. |
| | Indicator definition: Proportion of subjects with toxicity of grade 4 and 5 during |
| | the trial cycle. |
| | Evaluation methodology: Investigators recorded AEs that occurred during the |
| | clinical trial cycle and graded them according to CTCAE V5.0. |
| | (1) Objective Response Rate (ORR) (1 month± 7 days, 3 months, ± 7 days after the |
| | end of the last treatment). |
| | (2) Duration of Response (DOR) (3 months $\pm 7$ days) after the end of the last |
| | treatment |
| Secondary | (3) DCR (1 month $\pm 7$ days after the end of the last treatment). |
| effectiveness | (4) Tumor markers (if required) (screening period, 1 month $\pm 7$ days, 2 months $\pm 7$ |
| Evaluation | days, 3 months |
| indicators | (5) Tumor-specific symptoms (screening period, 1 month $\pm$ 7 days, 2 mon ths $\pm$ 7 days, |
| | 3 months ≠ days). |
| | (6) Product usability evaluation (ProBeam system, radiotherapy management software |
| | (OIS), radiotherapy planning software (Eclipse)) (the day of completion of the last |
| | treatment). |

- (1) CTCAE grade 1 and 2 toxicity ratio (3 months  $\pm 7$  days after the end of the last treatment).
- (2) Laboratory tests [screening period, treatment period on the 1st day of each week (Monday to Sunday is considered as 1 calendar week, the day of the first treatment of each natural week) before treatment or -1 day, 3 days after the end of the last treatment, 1 Months #7 days, 2 months #7 days, 3 months #7 days].

#### Secondary safety Evaluation indicators

- (3) Eastern Cooperative Oncology Group (ECOG) physical status grading [screening period, treatment period 1st day of each week (Monday to Sunday is regarded as 1 natural week, On the day of the first treatment of each calendar week) before or -1 day before treatment, within 3 days after the end of the last treatment, 1 month±7 days, 2 months±7 days, 3 months±7 days].
- (4) Tumor recurrence rate (3 months  $\pm 7$  days after the end of the last treatment).
- (5) Incidence of adverse events (AEs) (3 months  $\pm 7$  days after the end of the last treatment).
- (6) The incidence of Serious Adverse Events (SAEs) (3 months  $\pm 7$  days after the end of the last treatment).
- (7) Incidence of device defects (after last treatment)

Inclusion Criteria (Major Criteria):

- (1)  $18 \leq age \leq 80$  years;
- (2) First-diagnosed patients with tumors of the nervous system, head and neck, chest, abdomen, spine, pelvic cavity, limbs, etc. by tissue/cell pathology;
- (3) ECOG physical condition is graded as 0 to 2;
- (4) Women of childbearing had negative results in the blood pregnancy test (Human Chorionic Gonadotropin, HCG) 7 days prior to the first treatment;
- (5) The subject or subject's guardian is able to understand the purpose of the study, demonstrate sufficient compliance with the protocol and sign informed consent form.

## Eligibility criteria

#### Exclusion Criteria (Major Criteria):

- (1) The subject with radiotherapy contraindications, including the known genetic tendencies that increase the sensitivity of normal tissue radiotherapy or the accompanying diseases that lead to hypersensitivity to radiotherapy;
- (2) The subject with other uncontrolled tumors except that to be treated according to medical history or the investigator's estimation, or with other malignant tumors within five years prior to enrollment;
- (3) Implanted pacemakers or other metal prosthesis within the scope of proton therapy;
- (4) Other situations that investigator determines not suitable for enrollment.

#### Specifications for the use of investigational medical device

All subjects used the investigational medical device: ProBeam for radiation therapy.

Statistical analysis with SAS 9.4 software.

All data are described statistically, including baseline data, all efficacy measures, and all safety data. The measurement data give the mean, standard deviation, minimum, maximum, median, 25th quantile and 75th quantile; The counting data gives the frequency and composition ratio.

#### Effectiveness analysis

DCR was calculated and the Clopper-Pearson method was used to calculate the 95% confidence interval for tumor disease control. ORR was calculated and the Clopper-Pearson method was used to calculate the objective response rate 95% confidence interval. Descriptive statistics on the percentage change from baseline of the measurable sum of the longest diameter (SLD). The Waterfall Chart was made by the maximum percentage reduction in SLD per participant compared to the screening period.

The *Kaplan-Meier* method was used to calculate the median duration of response, median progression-free survival, median survival, and overall survival, and plotted *K-M* curves (long-term follow-up data).

Statistical analysis

#### Safey analysis

Descriptive statistics were used to classify organ systems in MedDRA medical terms, and the incidence, occurrence, and severity of adverse events, adverse reactions, and serious adverse events were summarized.

Laboratory indicators, ECOG physical status grading and other safety-related indicators were compared and evaluated before and after treatment, and clinical evaluation [no clinical significance, clinically significant (tends to normal), clinically significant (tends to be abnormal), not checked], CTCAE grade evaluation before and after treatment cross-tab.

The central effect is considered in the analysis process, and the general linear model is used for the measurement data and CMH for the counting data.

The baseline data analysis was performed using the Full Analysis Set (FAS); Effectiveness analysis uses FAS and Per Protocol Set (PPS); Security analysis uses the Safety Set (SS).

### **Trial flowchart**



#### The body of the protocol

#### 1 Sponsor information

#### 1.1 Name of the sponsor

Varian Medical Systems Trading (Beijing) Co., Ltd

#### 1.2 Sponsor address

No. 8 Yuncheng Street, Beijing Economic and Technological Development Zone, Beijing, 2nd floor, area B, 3rd floor

#### 1.3 The name, address, contact information and relevant qualification documents of the agent

NA

#### 2 Purpose and content of clinical trial

#### 2.1 Objective

Clinical trial (screening-short-term follow-up): The data obtained by using Proton Beam equipment (ProBeam) for radiation therapy in tumor patients compared with the target value to evaluate the effectiveness and safety of ProBeam for radiation therapy in tumor patients to provide clinical basis for product registration application.

Long-term follow-up: The long-term efficacy and safety of ProBeam for radiation therapy in cancer patients were evaluated by using the long-term follow-up data of ProBeam for radiation therapy in cancer patients.

#### 2.2 content

This clinical trial is a prospective study, carried out in 2 clinical trial institutions, and 47 patients with tumors of the nervous system, head and neck, chest, abdomen, spine, pelvis, limbs and other tumors were selected as study subjects, all using investigational medical devices, and designed for a single group of target values. The research device involved in this trial is the proton therapy device (ProBeam), a medical device for investigation. Short-term follow-up is: 1 visit during the screening period (within 4 weeks before the first treatment), 2~9 visits during the treatment period according to the length of treatment weeks (1~8 weeks), and 3 after the last treatment 3 visits within a month; Long-term follow-up was 11 visits over a period of 3~5 months after the end of the last treatment. The main efficacy evaluation index was DCR 3 months after the end of the last treatment, and the main safety evaluation index was the proportion of CTCAE grade 3 toxicity in the entire short-term follow-up clinical trial cycle and CTCAE 4 in the entire short-term follow-up clinical trial cycle The proportion of grade 5 toxicity reactions, the collected data were analyzed and compared with the target values, and the effectiveness and safety of ProBeam in proton radiation therapy for patients with tumors such as nervous system, head and neck, chest, abdomen, spine, pelvis, and extremities were evaluated. Tumor remission, recurrence, survival, device-related adverse events and serious adverse events were summarized 6 months, 1 year, 2 years and 5 years after the last treatment. To assess the long-term efficacy and safety of ProBeam for radiation therapy in patients with oncology.

#### 3 Overall design

#### 3.1 Trial design

#### 3.1.1 Trial and long-term follow-up purposes

#### 3.1.1.1 Main purpose

To evaluate whether the main efficacy evaluation index of ProBeam in radiotherapy for cancer patients reached the target value 3 months after the end of the last treatment. The main safety evaluation index: whether the proportion of CTCAE grade 3 toxicity is lower than the acceptable value, and whether CTCAE grade 4 and 5 toxic reactions occur.

#### 3.1.1.2 Secondary purposes

When evaluating the use of ProBeam in radiation therapy for tumor patients, the secondary effectiveness evaluation indicators ORR, DOR, DCR, tumor markers (if necessary), tumor-specific symptoms, and product usability evaluation are actually the actual situation.

When evaluating the use of ProBeam in radiation therapy in tumor patients, the proportion of secondary safety evaluation indicators CTCAE grade 1 and 2 toxicity, laboratory tests, ECOG physical status grade, tumor recurrence rate, adverse event rate, serious adverse event rate, The actual situation of the incidence of device defects.

#### 3.1.1.3 Long-term follow-up purposes

To evaluate the effectiveness of ProBeam for radiotherapy in tumor patients, the evaluation indexes were 6 months, 1 year, 2 years, 5 years of DCR The actual situation of ORR, DOR, PFS, OS.

After ProBeam was used in radiotherapy for tumor patients, the safety evaluation index was 6 months, 1 year, 2 years, and 5 years of device-related AE and device-related treatment SAE, the actual situation of tumor recurrence rate.

#### 3.1.2 Choice of trial method and justification

This trial was designed using the prospective, two-center, single-group target value method.

- (1) Prospective study: Adopt a research approach that traces from the present to the future. Prospective studies can establish cause and effect; There are unified diagnosis, detection and evaluation standards for the obtained data, so the data processing is controllable.
- (2) Two centers: Select 2 clinical trial institutions to carry out the clinical trial. More cases than single-center trials can be obtained in the same amount of time, thus shortening the duration of clinical trials.
- (3) Single-group target value method: Because the same device of the experimental medical device is radioactive and difficult to obtain, the existing treatment method is not feasible due to objective conditions, so the single-group target value method is adopted. Moreover, the applicable population and main evaluation indicators of experimental medical devices can be fully defined and relatively stable; The main evaluation index adopts the effective rate mentioned in the "Guidelines for the Technical Review of Clinical Evaluation of Proton Carbon Ion Therapy System" (CFDA Circular No. 4 [2018]), which is relatively objective and reproducible. According to the Guidelines for the Technical Review of Clinical Evaluation of Proton Carbon Ion Therapy Systems, the target value of therapeutic response rate for experimental medical devices should be at least 80%, and the expected value should be 95%. Among them, the effective definition is: CR+PR+SD (complete response CR, partial response PR, disease stable SD), which is basically consistent with the definition of tumor disease control rate in this clinical trial. Therefore, no control group was set up in this clinical trial, and the single-group target value method was used to evaluate whether the tumor disease control rate reached the target value (80%) and the main safety evaluation index CTCAE 3 when ProBeam was used in

radiotherapy for tumor patients Whether the proportion of grade toxicities is less than acceptable (5%) and whether the proportion of CTCAE grade 4 and 5 toxicities is acceptable (0%).

#### 3.1.3 Diagnostic and therapeutic methods of medical devices for investigation

All subjects used ProBeam, an investigational medical device. The investigator formulated an individualized radiotherapy plan according to the actual clinical situation of the subjects, and the use of experimental medical devices is detailed in the product manual.

The specific treatment process is: preoperative assessment to determine the indications (radiotherapist)  $\rightarrow$  signing of the informed consent form for radiotherapy (radiotherapist)  $\rightarrow$  selection and production of postural immobilization devices (radiotherapist, radiotherapist, physicist)  $\rightarrow$  CT/MRI Simulation positioning (radiotherapist, radiotherapist, physicist)  $\rightarrow$  target and normal organ delineation (radiotherapist)  $\rightarrow$  radiotherapy plan design (physicist)  $\rightarrow$  radiotherapy plan review and authorization for executable plans (radiotherapist, physicist),  $\rightarrow$  treatment plan validation (physicist),  $\rightarrow$  proton radiation therapy (radiotherapist). First treatment, radiotherapist and physicist are present)  $\rightarrow$  post-treatment efficacy evaluation (radiotherapist, independent imaging review team)  $\rightarrow$  follow-up (radiotherapist).

Subjects will receive radiotherapy with reference to the dose and segmentation prescribed by the trial, and the expected radiotherapy cycle of each subject is 1~8 weeks.

#### 3.1.3.1 Enrollment time

The investigators obtained the informed consent of the participants and signed the ICF, which was then screened according to the inclusion criteria. If the patient meets all the inclusion criteria of this trial and does not meet any of the exclusion criteria,

the case is included in this trial, and the time of enrollment of the subject is used as the treatment on the day of the first treatment, and a unique enrollment number is obtained in the order of enrollment.

#### 3.1.3.2 The number of subjects required for the clinical trial

After screening according to the inclusion criteria, it is expected that a total of 47 subjects will be included in this clinical trial, all of whom will be treated with investigational medical devices.

#### 3.1.4 Effectiveness evaluation methods

If it is not possible to follow up at the clinical trial center according to the visit arrangement due to the epidemic, the clinical examination can be examined by other tertiary hospitals, and the test results will be transmitted back to the clinical trial center for evaluation; The carrier of imaging data in the outer hospital is not limited, and it is necessary to ensure that the imaging department of the center can be opened and read.

## 3.1.4.1 The main effectiveness evaluation indicators and the methods and time selection of their evaluation, recording and analysis

(1) Tumor disease control rate (DCR).

Reason for selection: According to the clinical trial effectiveness evaluation in the "Guidelines for the Review of Clinical Evaluation Technologies of Proton Carbon Ion Therapy System" (CFDA Circular No. 4 [2018]): "In view of the local characteristics of radiotherapy, it is recommended that the efficacy evaluation should be based on local control, and according to the different diseases, the common standards in clinical research, such as the efficacy evaluation criteria for solid tumors, should be reasonably adopted RECIST. The efficacy evaluation can be divided into complete response CR, partial response PR, disease stable SD, disease progression PD, and the effective definition is: "CR+PR+SD." "; Due to the particularity of the disease, the evaluation method recommended in the relevant diagnosis and treatment guidelines is selected. The tumor disease

control rate was selected as the main effectiveness evaluation index, which was relatively objective and reproducible, and adopted the common standard in clinical research, which was widely recognized and applied by clinicians.

Definition of indicators: the occurrence of CR, PR and SD after the end of treatment is disease control; No biochemical recurrence at the end of prostate cancer treatment, no regional lymph nodes or distant metastases, considered disease control. Proportion of participants who developed disease control three months after the end of the last radiotherapy.

Metric type: Qualitative.

Data collection time: screening period, 3 months  $\pm$  7 days after the end of the last treatment.

Evaluation time: 3 months  $\pm$  7 days after the end of the last treatment.

Site of evaluation: Tumor receiving radiation therapy.

Evaluation method: The changes in tumor CT or MRI imaging before and after treatment were evaluated by an independent imaging review panel according to RECIST 1.1. At 3 months of radiographic evaluation, if PD is found, PET-CT is required to confirm it.

Calculation formula: DCR = number of disease control subjects / total number of subjects × 100%.

Criteria: See RECIST 1.1 for details. At the time of 3-month imaging evaluation, if the patient is found to have PD, PET-CT examination is required to confirm it, if progress is confirmed, it is recorded as PD, if progress cannot be confirmed, it may be false progression, and it is recorded as SD. If prostate cancer does not have biochemical recurrence, PET-CT examination is not required, and there is no metastasis by default, which is regarded as tumor control, and if biochemical recurrence occurs, it is regarded as tumor not controlled, and PET-CT is required to confirm tumor metastasis.

Note: Participants who aborted the trial for any reason (except loss to follow-up) before the end of the last radiation therapy were considered to have disease progression (PD) or were not controlled. Disease site evaluation uses the same approach as baseline, including consistent contrasted/non-contrast scans and prompt scanning. If changes are needed, the case must be discussed with a radiologist to determine whether an alternative approach is possible. If not, the objective situation in the future is unclear.

#### 3.1.4.2 Secondary effectiveness evaluation indicators and their methods and timing of evaluation, recording, analysis

(1) Objective response rate (ORR).

Reason for selection: The Guidelines for the Review of Clinical Evaluation Technologies of Proton Carbon Ion Therapy Systems (CFDA Circular No. 4 [2018]) recommends the use of the latest version of the commonly used evaluation criteria for radiation oncology as the clinical trial evaluation criteria, so RECIST 1.1 is used Relevant indicators as effectiveness evaluation criteria; Due to the particularity of the disease, the evaluation method recommended in the relevant diagnosis and treatment guidelines is selected. All of them can directly measure the effect of radiotherapy and are widely recognized and applied by clinicians.

Definition of indicators: CR or PR after the end of treatment is considered objective remission, prostate cancer has no biochemical recurrence at the end of the last treatment, and no regional lymph nodes or distant metastasis are considered objective remission. Proportion of participants who experienced objective remission at each time point after the end of the last treatment.

Metric type: Qualitative.

Data collection time: screening period, 1 month  $\pm$  7 days, 3 months,  $\pm$  7 days after the end of the last treatment.

Evaluation time: 1 month $\pm$  7 days, 3 months,  $\pm$  7 days after the last treatment.

Site of evaluation: Tumor receiving radiation therapy.

Evaluation method: The changes in tumor CT or MRI imaging before and after treatment were evaluated by an independent imaging review panel according to RECIST 1.1. At 3 months of radiographic evaluation, if PD is found, PET-CT is required to confirm it.

Calculation formula: ORR = number of subjects in objective response / total number of subjects  $\times$  100%.

Criteria: See RECIST 1.1 for details. At the time of 3-month imaging evaluation, if the patient is found to have PD, PET-CT examination is required to confirm it, if progress is confirmed, it is recorded as PD, if progress cannot be confirmed, it may be false progression, and it is recorded as SD. If prostate cancer does not have biochemical recurrence, PET-CT examination is not required, and there is no metastasis by default, which is regarded as objective remission, and if biochemical recurrence occurs, it is regarded as not objectively remission, and PET-CT is required to confirm tumor metastasis.

Note: Participants who aborted the trial for any reason (other than loss to follow-up) before the end of the last radiotherapy were considered to have not responded objectively. Disease site evaluation uses the same approach as baseline, including consistent contrasted/non-contrast scans and prompt scanning. If changes are needed, the case must be discussed with a radiologist to determine whether an alternative approach is possible. If not, the objective situation in the future is unclear.

#### (2) Time to sustained remission (DOR).

Reason for selection: The Guidelines for the Review of Clinical Evaluation Technologies of Proton Carbon Ion Therapy Systems (CFDA Circular No. 4 [2018]) recommends the use of the latest version of the commonly used evaluation criteria for radiation oncology as the clinical trial evaluation criteria, so RECIST 1.1 is used Relevant indicators as effectiveness evaluation criteria; Due to the particularity of the disease, the evaluation method recommended in the relevant diagnosis and treatment

guidelines is selected. They are all commonly used indicators for the evaluation of tumor treatment effects, and are widely recognized and applied by clinicians.

Indicator definition: the time between the first assessment of the tumour as CR or PR and the time between the first assessment of PD or death from any cause.

Indicator type: quantitative.

Data collection time: 1 month $\pm$  7 days, 3 months,  $\pm$  7 days after the end of the screening period, until tumor progression or subject death.

Evaluation time: 3 months  $\pm$  7 days after the last treatment.

Site of evaluation: Tumor receiving radiation therapy.

Evaluation method: The changes in tumor CT or MRI imaging before and after treatment were evaluated by an independent imaging review panel according to RECIST 1.1. At 3 months of radiographic evaluation, if PD is found, PET-CT is required to confirm it.

Calculation formula: DOR = time to death from PD or any cause on the first assessment - time to CR or PR for the first assessment;

Criteria: See RECIST 1.1 for details. At the time of 3-month imaging evaluation, if the patient is found to have PD, PET-CT examination is required to confirm it, if progress is confirmed, it is recorded as PD, if progress cannot be confirmed, it may be false progression, and it is recorded as SD.

Note: If no tumor progression or death is observed during the follow-up period after the end of radiotherapy, the formula is: DOR > last visit time after the end of the last radiotherapy - CR or PR time for first assessment. Others are the same as ORR.

(3) Tumor disease control rate (DCR).

Reason for selection: DCR 3 months after the end of the last treatment was the primary evaluation index, and DCR at other follow-up time was used as a secondary evaluation index.

Definition of indicators: the occurrence of CR, PR and SD after the end of treatment is disease control; No biochemical recurrence at the end of prostate cancer treatment, no regional lymph nodes or distant metastases, considered disease control. Proportion of participants who developed disease control at one month after the end of the last treatment.

Metric type: Qualitative.

Data collection time: screening period, 1 month  $\pm$  7 days after the end of the last treatment.

Evaluation time: 1 month  $\pm$  7 days after the last treatment.

Site of evaluation: Tumor receiving radiation therapy.

Evaluation method: The changes in tumor CT or MRI imaging before and after treatment were evaluated by an independent imaging review panel according to RECIST 1.1. At 3 months of radiographic evaluation, if PD is found, PET-CT is required to confirm it.

Calculation formula: DCR = number of disease control subjects / total number of subjects × 100%.

Criteria: See RECIST 1.1 for details. At the time of 3-month imaging evaluation, if the patient is found to have PD, PET-CT examination is required to confirm it, if progress is confirmed, it is recorded as PD, if progress cannot be confirmed, it may be false progression, and it is recorded as SD. If prostate cancer does not have biochemical recurrence, PET-CT examination is not required, and there is no metastasis by default, which is regarded as tumor control, and if biochemical recurrence occurs, it is regarded as tumor not controlled, and PET-CT is required to confirm tumor metastasis.

Note: Participants who aborted the trial for any reason (other than loss to follow-up) before the end of the last radiotherapy were considered to have PD or was uncontrolled. Disease site evaluation uses the same approach as baseline, including consistent contrasted/non-contrast scans and prompt scanning. If changes are needed, the case must be discussed with a radiologist to determine whether an alternative approach is possible. If not, the objective situation in the future is unclear.

#### (4) Tumor markers (if needed)

Reason for selection: The Guidelines for the Review of Clinical Evaluation Technologies of Proton Carbon Ion Therapy System (CFDA Circular No. 4, 2018) suggests that changes in tumor markers and functional imaging parameters should be used as reference factors for effectiveness evaluation.

Data collection and evaluation time: screening period, 1 month  $\pm$  7 days, 2 months $\pm$  7 days, 3 months $\pm$  7 months after the end of the last treatment Sky.

Evaluation method: tumor marker examination is performed, and the investigator judges that the tumor marker (before and after radiotherapy) is reported as clinically significant changes.

Note: Researchers choose relevant indicators according to the disease, and the scheme is not uniformly stipulated.

#### (5) Tumor-specific symptoms

Reason for selection: The Guidelines for the Review of Clinical Evaluation Technologies of Proton Carbon Ion Therapy Systems (CFDA Circular No. 4 of 2018) suggests that clinical manifestations should be recorded during follow-up.

Data collection and evaluation time: screening period, 1 month  $\pm$  7 days, 2 months $\pm$  7 days, 3 months $\pm$  7 months after the end of the last treatment Sky.

Methodology: Symptoms are recorded according to the type of disease, which may include, but are not limited to, the following: pain, swallowing function, mobility, bleeding, visual acuity, appetite/weight, superficial lymph node size, and the investigator judges that the symptoms (before and after radiotherapy) are clinically significant.

Note: Researchers record relevant symptoms according to the disease, and the plan is not uniformly stipulated.

(6) Product usability evaluation (ProBeam system, radiotherapy management software (OIS), radiotherapy planning software (Eclipse)).

Reason for selection: Routine effectiveness indicators of medical device clinical trials.

Indicator type: quantitative, open-ended question.

Data collection and evaluation time: the day the last treatment was completed.

Evaluation method: Researchers using the corresponding function scored according to the Likrt scale and collected openended questions to evaluate the overall feeling of ease of use during treatment.

#### 3.1.5 Safety evaluation methods

If it is not possible to follow up at the clinical trial center according to the visit arrangement due to the epidemic, the clinical examination can be examined by other tertiary hospitals, and the test results will be transmitted back to the clinical trial center for evaluation; The carrier of imaging data in the outer hospital is not limited, and it is necessary to ensure that the imaging department of the center can be opened and read.

## 3.1.5.1 The main safety evaluation indicators and the methods and time selection of their evaluation, recording and analysis

#### (1) CTCAE 3 toxicity ratio

Reason for selection: According to the Guidelines for the Technical Review of Clinical Evaluation of Proton Carbon Ion Therapy System (CFDA Circular No. 4 of 2018), if the proportion of CTCAE grade 3 acute toxic reactions exceeds 5%, it is considered as a clinical trial failure, so it is selected. The proportion of CTCAE grade 3 toxicity is used as the main safety evaluation index, and CTCAE is a commonly used safety evaluation standard in radiation oncology, which is widely recognized and applied by clinicians.

Indicator definition: Proportion of subjects with grade 3 toxicity during the trial cycle.

Metric type: Qualitative.

Data collection time: the entire clinical trial cycle.

Evaluation time: 3 months  $\pm$  7 days after the last treatment.

Evaluation methodology: Investigators recorded AEs that occurred during the clinical trial cycle and graded them according to CTCAE V5.0.

Calculation formula: proportion of CTCAE grade 3 toxicities = (number of subjects with CTCAE grade 3 toxicity in the test cycle) / total number of subjects  $\times$  100%.

Judging criteria: See CTCAE V5.0 for details.

(2) CTCAE Grade 4 and 5 toxicity ratio

Reason for selection: According to the Guidelines for the Review of Clinical Evaluation Technologies of Proton Carbon Ion Therapy System (CFDA Circular No. 4 of 2018), CTCAE grade 4 and 5 toxicities are considered to be clinical trial failures, so 4 is selected. The proportion of grade 5 and grade 5 toxicity reactions is used as a safety evaluation index, and CTCAE is a commonly used safety evaluation standard in radiation oncology, which is widely recognized and applied by clinicians.

Indicator definition: Proportion of subjects with toxicity of grade 4 and 5 during the trial cycle.

Metric type: Qualitative.

Data collection time: the entire clinical trial cycle.

Evaluation time: 3 months  $\pm$  7 days after the last treatment.

Evaluation methodology: Investigators recorded AEs that occurred during the clinical trial cycle and graded them according to CTCAE V5.0.

Formula: Proportion of CTCAE grade 4 and 5 toxicities = (number of subjects with CTCAE grade 4 and 5 reactions in the test cycle) / total number of subjects  $\times$  100%

Judging criteria: See CTCAE V5.0 for details.

#### 3.1.5.2 Secondary safety evaluation indicators and their methods and time selection for evaluation, recording and analysis

#### (1) CTCAE grade 1 and 2 toxicity ratio

Reason for selection: The proportion of CTCAE grade 3~5 toxicity reactions 3 months after the end of the last treatment was the main safety evaluation index, and the proportion of CTCAE grade 1 and grade 2 toxicity reactions was used as a secondary safety evaluation index for auxiliary evaluation.

Indicator definition: Proportion of subjects with grade 1 and 2 toxicity during the trial cycle.

Metric type: Qualitative.

Data collection time: the entire clinical trial cycle.

Evaluation time: 3 months  $\pm$  7 days after the last treatment.

Evaluation methodology: Investigators recorded AEs that occurred during the clinical trial cycle and graded them according to CTCAE V5.0.

Calculation formula: proportion of CTCAE grade 1 and 2 toxicities = (number of subjects with CTCAE grade 1 and 2 toxicities in the test cycle) / Total number of participants× 100%.

Judging criteria: See CTCAE V5.0 for details.

#### (2) Laboratory tests

Reason for selection: According to the Guidelines for Technical Review of Clinical Evaluation of Proton Carbon Ion Therapy System (CFDA Circular No. 4 of 2018), changes in clinical symptoms and signs should be recorded for clinical manifestations, tumor improvement (imaging examinations, laboratory test data), etc., and comprehensive analysis should be carried out. At the same time, it is a routine safety monitoring index for medical device clinical trials.

Data collection and evaluation time: screening period, treatment period 1st day per week (Monday to Sunday is regarded as 1 calendar week, each natural week on the day of the first treatment), before treatment or -1 day (blood count only), 3 days after the end of the last treatment, 1 month  $\pm$  7 days (except coagulation routine), 2 months $\pm$  7 days (except coagulation routine).  $\odot$ 

Evaluation items: blood routine, coagulation routine, urine routine, liver function, kidney function.

Evaluation method: Laboratory tests are performed and the investigator judges clinically significant changes in laboratory indicators (before and after radiotherapy).

#### (3) ECOG grading of physical status

Reason for selection: According to the Guidelines for the Review of Clinical Evaluation Technologies of Proton Carbon Ion Therapy System (CFDA Circular No. 4 of 2018), the follow-up of subjects should include safety and efficacy evaluation. The general condition of the subjects is recommended to be evaluated using the internationally accepted scoring method.

Data collection time and evaluation time: screening period, treatment period on the first day of each week (every Monday to Sunday is regarded as 1 calendar week, each natural week on the day of the first treatment) before treatment or -1 day, 3 days after the end of the last treatment, 1 month  $\pm$  7 days, 2 months $\pm$  7 days, 3 months,  $\pm$  7 days.

Evaluation method: ECOG physical performance status was graded and reported by the investigator to report clinically significant changes in the test results (before and after radiotherapy).

#### (4) Tumor recurrence rate

Reason for selection: According to the Guidelines for the Review of Clinical Evaluation Technologies of Proton Carbon Ion Therapy System (CFDA Circular No. 4 of 2018), the clinical trial summary report still needs to be submitted 6 months, 1 year and 2 months after treatment. The situation in years and 5 years is summarized, including the tumor recurrence rate. Therefore, an adjuvant analysis of tumor recurrence rate was also added to short-term follow-up. At the same time, it is a common indicator for the safety evaluation of tumor treatment, and is widely recognized and applied by clinicians.

Definition of indicators: The tumor recurrence rate is the ratio of the number of subjects with tumor recurrence to the total number of subjects. Tumor recurrence refers to tumors that are clinically controlled after radiation therapy and regrow after a period of time, in the same nature as the primary tumor. Clinically referred to recurrence mostly refers to local recurrence, such as remnant organs, irradiation fields, and affected adjacent organs. Prostate cancer recurrence refers to biochemical recurrence and PET-CT is required to confirm tumor metastasis to lymph nodes or distant metastases.

Metric type: Qualitative.

Data collection time: screening period, 1 month $\pm$  7 days, 3 months,  $\pm$  7 days after the last treatment.

Evaluation time: 3 months  $\pm$  7 days after the last treatment.

Evaluation method: The changes in tumor CT or MRI imaging before and after treatment were evaluated by an independent imaging review panel according to RECIST 1.1. At 3 months of radiographic evaluation, if PD is found, PET-CT is required to confirm it.

Calculation formula: tumor recurrence rate = number of subjects with tumor recurrence / total number of subjects × 100%.

Criteria: See RECIST 1.1 for details. At the time of 3-month imaging evaluation, if the patient is found to have PD, PET-CT examination is required to confirm it, if progress is confirmed, it is recorded as PD, if progress cannot be confirmed, it may be false progression, and it is recorded as SD. If prostate cancer does not have biochemical recurrence, PET-CT examination is not required, and there is no metastasis by default, which is regarded as tumor control, and if biochemical recurrence occurs, it is regarded as tumor not controlled, and PET-CT is required to confirm tumor metastasis.

Note: Participants who discontinued the trial for any reason (other than loss to follow-up) before the end of radiotherapy were considered to have no oncological disease control. Disease site evaluation uses the same approach as baseline, including

consistent contrasted/non-contrast scans and prompt scanning. If changes are needed, the case must be discussed with a radiologist to determine whether an alternative approach is possible. If not, the objective situation in the future is unclear.

#### (5) Adverse event rate

Reason for selection: Routine safety monitoring indicators for clinical trials of medical devices.

Indicator definition: Adverse events are adverse medical events that occur during clinical trials, whether or not related to a device.

Metric type: Qualitative.

Data collection time: the entire clinical trial cycle.

Evaluation time: 3 months  $\pm$  7 days after the last treatment.

Evaluation method: The investigator recorded all AEs that occurred.

Calculation formula: adverse event rate = number of subjects with adverse events in this group / total number of subjects in this group  $\times$  100%.

#### (6) Serious adverse event rate

Reason for selection: Routine safety monitoring indicators for clinical trials of medical devices.

Definition: Serious adverse events are those that occur in the course of a clinical trial that result in death or serious deterioration of health, including fatal illness or injury, permanent defects in body structure or function, requiring hospitalization or prolonged hospital stay, or requiring medical or surgical intervention to avoid permanent defects in body structure or body function; Events that lead to fetal distress, fetal death, or congenital anomalies or birth defects.

Metric type: Qualitative.

Data collection time: the entire clinical trial cycle.

Evaluation time: 3 months  $\pm$  7 days after the last treatment.

Evaluation methodology: The investigator recorded all SAEs that occurred.

Calculation formula: Serious adverse event rate = number of subjects with serious adverse events in this group / total number of subjects in this group  $\times$  100%.

#### (7) Incidence of device defects

Reason for selection: Routine safety monitoring indicators for clinical trials of medical devices.

Definition of indicators: refers to the unreasonable risk that medical devices may endanger human health and life safety under normal use during clinical trials, such as crash.

Metric type: Qualitative.

Time of data collection: during treatment.

Evaluation time: After the last treatment was completed.

Evaluation methodology: The investigator recorded all device defects that occurred.

Calculation formula: incidence of device defects = number of occurrences of device defects / number of times of device use  $\times$  100%.

#### 4 Statistical considerations

#### 4.1 Statistical design, methods, and analytical protocols

This study was a prospective, two-center, single-group target value trial.

All statistical analysis methods are described in detail in the statistical analysis plan. A first draft of the statistical analysis plan is formed after the protocol and eCRF are finalized and will be finalized prior to database locking.

#### 4.2 Sample size calculation

#### 4.2.1 Total sample size

This clinical trial intends to enroll 47 subjects. The sample size determination process is as follows:

This clinical study is designed for clinical verification of a single group of target values, and the tumor disease control rate, the main effectiveness evaluation index, is used as the basis for sample size estimation. According to the Guidelines for the Review of Clinical Evaluation Technologies of Proton Carbon Ion Therapy System (CFDA Circular No. 4 of 2018), the target value is set at 80%, and the bilateral significance level is 0.05, and the power degree 80%, applying the sample size estimation professional software PASS 15.0, calculated by the above parameters, the test group needs a sample size of at least 42 cases. Considering that about 10% of cases may be dropped or lost to follow-up during clinical validation, the sample size of the experimental group was expanded to 47 cases.

#### 4.3 The level of significance and power of clinical trials

The significance level  $\alpha$  (bilateral) = 0.05, and the power was 80%.

#### 4.4 Expected shedding rate

In the sample size estimation process, the expected shedding rate is 10%.

This dropout rate refers to the proportion of participants who ultimately could not be included in the primary analysis. Shedding subjects are subjects who have been identified by the investigator as having serious protocol deviations. May include, but is not limited to, the following: the subject violates the inclusion criteria; Participants were not treated with experimental devices; Participants used concomitant medications/devices that are prohibited by the protocol; lack of data on key evaluation indicators; Participants did not obtain any data, etc.

#### 4.5 Criteria for passing/failing clinical trial results

The target value of the main effectiveness evaluation index (tumor disease control rate) of the trial was 80%, and if the lower limit of the 95% confidence interval of the test results was greater than 80%, the tumor disease control rate of the experimental group reached the target.

If the main safety evaluation index of the trial (the proportion of CTCAE grade 3 toxic reactions) is greater than 5%, the clinical trial fails.

If the trial has CTCAE grade 4 and 5 toxicity, the clinical trial fails.

#### 4.6 Criteria and reasons for terminating trials on statistical grounds

No interim analysis was performed in this study and therefore criteria for termination of the trial for statistical reasons were not established.

# 4.7 Statistical methods of data, together with methods of dealing with missing, unused or erroneous data and irrational data

#### 4.7.1 Data statistical methods

Statistical analysis with SAS 9.4 software.

All data are described statistically, including demographics, baselines, all efficacy measures, and all safety data. The measurement data give the mean, standard deviation, minimum, maximum, median, 25th quantile and 75th quantile; The counting data gives the frequency and the corresponding percentage.

Effectiveness Analysis:

The number and percentage of cases achieving DCR were calculated, and the Clopper-Pearson method was used to calculate the 95% confidence interval for tumor disease control rate. ORR was calculated and the Clopper-Pearson method was used to calculate the objective response rate 95% confidence interval. Descriptive statistics on the percentage change from baseline of the sum of the longest diameter (SLD) of the measurable tumor. The Waterfall Chart was made by the maximum percentage reduction in SLD per patient compared to the screening period.

The *Kaplan-Meier* method was used to calculate the median duration of response, median progression-free survival, median survival, and overall survival, and plotted *K-M* curves (long-term follow-up data).

For tumor markers, compare and evaluate the changes before and after treatment, and give clinical evaluation [no clinical significance, clinically significant (tend to normal), clinically significant (tend to be abnormal), not checked].

Safety Analysis:

Descriptive statistics were used to classify organ systems in MedDRA medical terms, and the incidence, occurrence, and severity of adverse events, adverse reactions, and serious adverse events were summarized.

Laboratory indicators, ECOG physical status classification and other safety-related indicators were compared and evaluated before and after treatment, and clinical evaluation ([no clinical significance, clinically significant (tending to normal), clinically significant (tending to abnormal), not checked], CTCAE grade evaluation before and after treatment cross-table.

# 4.7.2 Missing, unused, or erroneous data (including mid-exit and evacuation) and unreasonable data

All missing, unused or erroneous data (including mid-exit and withdrawal) and unreasonable data will be discussed and finalized by investigators and

biostatisticians during the blinding review phase. The basic statistical principles of these data processing are as follows:

- (1) Describe the details of each shedding case;
- (2) Missing data from baseline, which can not be estimated;
- (3) The missing values of DCR and primary safety evaluation indicators (proportion of CTCAE grade 3 toxicities, proportion of CTCAE grade 4 and 5 toxicities) at 3 months after the end of treatment can be estimated using worst-case scenarios.
- (4) The missing values of qualitative secondary effectiveness evaluation indicators ORR, DCR and long-term follow-up effectiveness evaluation indicators can be estimated using worst-case scenarios;
- (5) The missing values of quantitative secondary efficacy evaluation indicators DOR, tumor markers, product ease assessment and long-term follow-up effectiveness evaluation indicators were not estimated.
- (6) Erroneous, unreasonable data (out-of-range data and data that contradicts other data or indicators of the study protocol) can be treated as missing values;
- (7) Worst-case estimates are used for missing values for all minor safety indicators;

- (8) The sensitivity analysis of the main effectiveness evaluation indicators and main safety evaluation indicators after treatment was carried out in the whole analysis center.
- (9) The sensitivity analysis of all secondary effectiveness evaluation indicators after treatment was carried out in the whole analysis center.
- (10) For all secondary safety evaluation indicators after treatment, sensitivity analysis was carried out in the security dataset.

#### 4.8 Procedures for reporting deviations from the original statistical plan

Under normal circumstances, only the statistical analysis content agreed in advance included in the statistical analysis plan can be presented in the clinical trial report of this trial. The increased demand for statistical analysis for various uncertain reasons is only exploratory analysis.

#### 4.9 Selection criteria and rationale for participants included in the analysis

Full Analysis Set (FAS): All subjects who received at least 1 investigational device treatment and at least one post-baseline observation data will be enrolled in FAS, according to the basic principles of intention-to-heart analysis. FAS will be used as the primary population for baseline data and sensitivity analysis for validity evaluation. Participants may only be excluded in very limited circumstances, including when important inclusion criteria are violated and no observational data are available after enrollment.

Compliant protocol set (PPS): is a subset of FAS, defined as subjects who have measurable lesions at baseline and have completed at least one assessment of primary efficacy indicators after baseline. PPS will be the primary population for the effectiveness evaluation of this study.

Safety dataset (SS): all participants who received at least 1 study device treatment and at least one safety assessment. SS will be the primary population for safety analysis in this study.

The assessment of baseline characteristics will use the full set of analyses;

The evaluation of effectiveness will use both the full analysis set and the
conforming protocol set; Security analysis uses security datasets.

#### 4.10 Covariate and subgroup analysis

Subgroup analysis as necessary was not precluded. Subgroups include, but are not limited to:

(1) Tumor sites (tumors of the nervous system, head and neck, chest, abdomen, spine, pelvis, extremities, etc.).